CLINICAL TRIAL: NCT03612167
Title: Constructing A Model of Health Promotion and Active Aging for Community-Dwelling Older Adults
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: no funding
Sponsor: National Cheng Kung University (Other)
Collaborators: Chang Gung University of Science and Technology (Other)
Responsible Party: Principal Investigator, Ling-Hui Chang, Associate Professor, National Cheng Kung University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 102-2717B
Record Dates: First submitted 2018-07-22; First posted 2018-08-02 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Subjective Cognitive Complaints

STUDY DESIGN:
Intervention Model Description: A quasi-experimental design with nonequivalent control was adopted in a senior center. Experimental variable was a 12 consecutive 90-minute weekly cognitive groups that included cognitive training and rehabilitation, with activity-based cognitive exercises and discussions with a focus on applications of cognitive strategies in daily lives. Participants were allocated into intervention group (cognitive intervention group) and control group (nutrition education group). The group assignment depended on what group they signed up for participate.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- multi-modal cognitive intervention (Experimental): a 12 consecutive 90-minute weekly cognitive groups that included cognitive training and rehabilitation, with activity-based cognitive exercises and discussions with a focus on applications of cognitive strategies in daily lives.
  Interventions: Behavioral: cognitive intervention
- nutritional group (Active Comparator): A quasi-experimental design with nonequivalent control was adopted in a senior center. The intervention for control group was a 12 consecutive 90-minute weekly nutritional groups that included nutrition classes (lecture and discussion).
  Interventions: Behavioral: nutritional group

INTERVENTIONS:
Behavioral: cognitive intervention — a 12 consecutive 90-minute weekly cognitive groups that included cognitive training and rehabilitation, with activity-based cognitive exercises and discussions with a focus on applications of cognitive strategies in daily lives.
  Arms: multi-modal cognitive intervention
Behavioral: nutritional group — 12 consecutive 90-minute weekly nutritional groups that included nutrition classes (lecture and discussion).
  Arms: nutritional group

SUMMARY:
Cognitive intervention for people with subjective cognitive complaints can be categorized into cognitive training, cognitive rehabilitation, psychoeducation, lifestyle intervention, etc. Literature have suggested multicomponent cognitive interventions can have better outcomes. However, studies to support this proposition are still limited. Few studies have also examined the influences of cognitive intervention on functional performance. This study was to examine the effectiveness of a multicomponent cognitive intervention for community-dwelling elderly with subjective cognitive complaints.

ELIGIBILITY:
Inclusion Criteria:

1. Subjective cognition complaint by the client or caregiver: In our study, participants reported more than one complaint in Everyday Memory Questionnaire and Cognitive Function Questionnaire will be included.
2. Objective cognition deficits: participants with scores under 1.5 Standard Deviation in Trail making test, Contextual memory test and Rivermead Behavior Memory Test-3rd edition were included.
3. Preserved most daily living function: participants have reported no Activity of Daily Living (ADL) difficulties.

Exclusion Criteria:

1. A confirmed diagnosis of dementia
2. With visual and auditory impairments, and other neurocognitive disease that can potential influence participation in group activities, including stroke, Parkinson's disease and traumatic brain injury, major depression, and substance abuse.
3. With Mini Mental Status Exam <=24 (education status beyond primary school); or <=16 (No education)
4. With less than 10-session participation rate out of 12.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2013-03-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
The Mini-Mental State Examination | 3 month
  cognition
the Trail Making Test | 3 month
  attention
the Color Trail Test | 3 month
  attention
Rivermead Behavioral Memory Test | 3 month
  memory
the Contextual Memory Test | 3 month
  memory
the Digit Span test | 3 month
  memory

SECONDARY OUTCOMES:
Cognitive Failure Questionnaire and the | 3 month
  perceived cognitive failures
Everyday Memory Questionnaire | 3 month
  perceived memory problems

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng-Kung University, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No
On-going research. Individual data will only share within the research team.